CLINICAL TRIAL: NCT03667287
Title: Full-thickness Skin vs. Synthetic Mesh in the Repair of Parastomal Hernia
Brief Title: Stoma Hernia Intraperitoneal Full-Thickness Skin
Acronym: SHIFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-251-31M
Record Dates: First submitted 2018-08-29; First posted 2018-09-12 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2018-08

CONDITIONS: Parastomal Hernia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full-thickness skin graft (Experimental): Repair of parastomal hernia with full-thickness skin graft, placed intraperitoneally, as reinforcement.
  Interventions: Procedure: Repair of parastomal hernia
- Synthethic mesh (Active Comparator): Repair of parastomal hernia with best available conventional method, using synthetic mesh material as reinforcement
  Interventions: Procedure: Repair of parastomal hernia

INTERVENTIONS:
Procedure: Repair of parastomal hernia — Surgical repair of symptomatic parastomal hernia.

SUMMARY:
This is a prospective randomized study to compare surgical methods for the repair of parastomal hernia.

DETAILED DESCRIPTION:
Parastomal hernia is a common complication to a stoma which can cause considerable suffering for the patient. The conventional methods of repair available today have disappointing results with high recurrence rates and serious complications. Some of the complications can be related to the introduction of foreign material into the abdominal wall. The investigators hypothesis is that the use of autologous full-thickness skin graft as reinforcement material can offer an alternative with fewer complications and recurrences.

Patients with symptomatic parastomal hernia will be included in a prospective randomized multicenter study comparing reinforcement with conventional synthetic mesh (with the best available technique today), to full thickness skin grafts placed in an intraperitoneal position. The intervention will be blinded to the participants, nursing staff and the follow-up staff. The participants will be followed up at 3, 12 and 36 months monitoring complications, recurrences, quality of life, strength of the abdomino-lumbar girdle and calculations will be done on the health economics.

ELIGIBILITY:
Inclusion Criteria:

* Colo-, ileo- or urostomy
* Parastomal hernia diagnosed with intrastomal ultrasound and/or CT
* Symptoms from the parastomal hernia requiring surgical intervention
* Informed consent
* >18 years of age
* Sufficient knowledge in the Swedish language so that questionnaires can be answered

Exclusion Criteria:

* Cognitive impairment unabling compliance to post-operative prescriptions and/or answering questionnaires
* Insufficient amount of good quality skin suitable for transplantation
* Expected high donor-site morbidity
* Fistula/e adjacent to stoma
* Mb Crohn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of complications at 3 months | 3 month post-operative clinical follow-up
  Complications will be assessed over a 3 year period of regular follow-up by an objective surgeon who is unaware of which surgical method which was used. Eventual complications may include infection, bleeding, seroma and fistula formation.

SECONDARY OUTCOMES:
Recurrence | 3, 12 and 36 months
  Parastomal hernia recurrence measured clinically, with stomal ultrasound and/or computerized tomography.
Pain - VHPQ | 3, 12 and 36 months.
  All subjects will complete Ventral Hernia Pain Questionaire (VHPQ) to assess and compare pre- and postoperative pain.
QoL - EORTC CR29 | 3, 12 and 36 months.
  All subject will complete European Organisation for Research and Treatment of Cancer questionnaire module for colorectal cancer (EORTC CR29) as a complement to EORTC C30, to assess and compare pre- and postoperative quality of life.
QoL - EORTC C30 | 3, 12 and 36 months.
  All subject will complete European Organisation for Research and Treatment of Cancer core quality of life questionnaire (EORTC CR30) to assess and compare pre- and postoperative quality of life.
Abdominal strength | 12 and 36 months.
  Strength of the abdomino-lumbar girdle measured in Biodex-4.
Health economics | 12 and 36 months.
  Cost-effectiveness of the separate procedures. The total cost of each method will be calculated from the hospital economic systems including duration of surgery, cost of operating time and equipment as well as duration and cost of anesthesia.
Rate of complications at 12 months | 12 month post-operative clinical follow-up
  Complications will be assessed over a 3 year period of regular follow-up by an objective surgeon who is unaware of which surgical method which was used. Eventual complications may include infection, bleeding, seroma and fistula formation.
Rate of complications at 36 months | 36 month post-operative clinical follow-up
  Complications will be assessed over a 3 year period of regular follow-up by an objective surgeon who is unaware of which surgical method which was used. Eventual complications may include infection, bleeding, seroma and fistula formation.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Strigård, PhD, Principal Investigator — Umeå University, Department of Surgical and Perioperative sciences
Locations (2):
- Sweden (2):
  - Sunderby Hospital, Luleå, Norrbotten County
  - University Hospital of Umeå, Umeå, Västerbotten County

REFERENCES:
- [Derived] Holmdahl V, Gunnarsson U, Strigard K. Autologous full-thickness skin graft as reinforcement in parastomal hernia repair: a randomised controlled trial. Trials. 2021 Dec 7;22(1):891. doi: 10.1186/s13063-021-05884-4. PMID 34876195